CLINICAL TRIAL: NCT00003985
Title: Phase I Study of KRN7000 in Patients With Solid Tumor Treated With a Weekly Intravenous Administration Schedule
Brief Title: KRN7000 in Treating Patients With Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-13972; EORTC-13972; KIRIN-EORTC-13972
Record Dates: First submitted 1999-11-01; First posted 2004-05-25 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: non-small cell lung cancer; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — KRN 7000

INTERVENTIONS:
Drug: KRN7000

SUMMARY:
RATIONALE: Biological therapies such as KRN7000 use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: Phase I trial to study the effectiveness of KRN7000 in treating patients who have solid tumors that have not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety profile and maximum tolerated dose of KRN7000 in patients with solid tumors. II. Assess the biological and immunological parameters that would suggest the optimal biologically active dose of KRN7000 in these patients. III. Determine the pharmacokinetics of KRN7000 at the different dose levels in these patients. IV. Measure any antitumor activity in these patients treated with this regimen.

OUTLINE: This is a dose escalation study. Patients receive KRN7000 by slow intravenous injection on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients each receive escalating doses of KRN7000 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which at least 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven solid tumor that is refractory to conventional treatment or for which no curative or standard palliative treatment exists No brain involvement or leptomeningeal disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG/WHO 0-2 Life expectancy: At least 3 months Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 100,000/mm3 Lymphocyte count at least 600/mm3 Hepatic: Bilirubin less than 1.5 mg/dL AST and ALT no greater than 2.5 times upper limit of normal No liver cirrhosis Hepatitis B surface antigen negative Renal: Creatinine no greater than 1.4 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No New York Heart Association class III or IV heart disease Immunologic: No immunodeficiency No autoimmune disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No active infection No nonmalignant disease incompatible with study No prior alcoholism, drug addiction, or psychotic disorders unless suitable for adequate follow up No cerebroside metabolite abnormalities (e.g., Gaucher's disease) HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 months since prior immunotherapy No concurrent cytokines Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas, mitomycin, and high dose chemotherapy) Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy (6 weeks for extensive radiotherapy) No concurrent radiotherapy Surgery: Not specified Other: No other concurrent investigational or antitumor drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1998-09

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, MD, PhD, Study Chair — Free University Medical Center
Locations (27):
- Austria (2):
  - Innsbruck Universitaetsklinik, Innsbruck
  - Kaiser Franz Josef Hospital, Vienna
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Ludwig Institute for Cancer Research-Brussels Branch, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Herlev Hospital - University Hospital of Copenhagen, Herlev, Denmark
- France (5):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Universitaetsklinik und Strahlenklinik - Essen, Essen
  - Klinikum Nurnberg, Nuremberg (Nurnberg)
- Netherlands (5):
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Ziekenhuis der Vrije Universiteit, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - University Medical Center Nijmegen, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
- Norwegian Radium Hospital, Oslo, Norway
- Switzerland (3):
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Kantonsspital - Saint Gallen, Sankt Gallen
- United Kingdom (4):
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - C.R.C. Beatson Laboratories, Glasgow, Scotland